CLINICAL TRIAL: NCT07056205
Title: Comparative Expression of ER,PR and HER2/Neu in Initial and Recurrent Breast Cancer.
Status: Enrolling by invitation | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Abdelmoaty Nafady Abdelmoaty, Comparative expression of ER, PR and HER2/neu in initial and recurrent breast cancer., Sohag University
Other Study IDs: Soh-Med--25-5-1MS
Record Dates: First submitted 2025-06-29; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
Keywords: ER,PR,HER2/neu,breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Archived histological slides and immune-stained slides of 100 patient with initial and recurrent mammary carcinoma will be obtained from Pathology Laboratory at Sohag Oncology Center.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- archived histological slides and immune-stained slides of 100 patient with breast cancer

SUMMARY:
Expression of ER, PR and HER2/neu in initial and recurrent breast cancer and correlate the results to different clinical and pathological parameters as patient age,sex, tumor location, status of nodal involvement and lymphovascular invasion

DETAILED DESCRIPTION:
Clinical data, pathological data, expression status of ER, PR and HER2/neu of both initial tumor and recurrent tumor and received treatment for BC patients diagnosed between January 2021 and December 2024 will be extracted from archive of multidisciplinary team (MDT) for management of BC at Sohag Oncology Center. In addition; hematoxylin and eosin stained slides and immune-stained slides for ER, PR and HER2/neu for selected patient's will be retrieved from archives of Pathology unit at Sohag Oncology Center and reviewed to confirm pathological features, ER expression, PR expression and HER2 status of both initial and recurrent tumor tissues.

ELIGIBILITY:
Inclusion Criteria:

Patients with excised breast cancer then experienced recurrence at same site. Patients with evaluated ER, PR and HER2/neu for both initial and recurrent tumors.

Exclusion Criteria:

* Cases with insufficient clinical of pathological data. Deficient ER, PR and HER2/neu status in either initial or recurrent tumor

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — - Inclusion criteria: Patients with excised breast cancer then experienced recurrence at same site. Patients with evaluated ER, PR and HER2/neu for both initial and recurrent tumors.
  - Exclusion criteria: Cases with insufficient clinical of pathological data. Deficient ER, PR and HER2/neu status in either initial or recurrent tumor
Study Population: archived histological slides and immune-stained slides of100 patient with initial and recurrent mammary carcinoma will be obtained from Pathology Laboratory at Sohag Oncology Center.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Comparison between initial and recurrent breast cancer in immunohistochemical expression of ER,PR and HER2/neu | 6 months

SECONDARY OUTCOMES:
Correlate the results of immunohistochemical expression of ER,PRand HER2/neu with the patients age ,sex,nodal status and lymphovascular invasion | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
No decided